CLINICAL TRIAL: NCT00002189
Title: Paclitaxel in Advanced Refractory Kaposi's Sarcoma (AIDS-KS): A Phase II Trial of Paclitaxel From Baker Norton Pharmaceuticals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baker Norton Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 273A; IX-110-081
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-06

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Paclitaxel; Treatment Outcome; Antineoplastic Agents, Phytogenic
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel

SUMMARY:
To determine response rate, median time to tumor progression, qualitative and quantitative toxicity and reversibility of toxicity in patients with advanced refractory AIDS-associated Kaposi's sarcoma (KS) administered a 3-hour infusion of paclitaxel every 14 days. To evaluate the clinical benefit of paclitaxel in this patient population by evaluating self-reported responses to the Symptom Distress Scale and by documenting and evaluating any changes in their lymphedema, pain and disfiguring facial lesions.

DETAILED DESCRIPTION:
Patients are treated with paclitaxel intravenously every 2 weeks up to 10 courses. Patients who achieve a complete response receive 2 additional courses those who achieve partial response or stabilization, continue therapy until progression.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Microscopically confirmed diagnosis of KS associated with HIV for which systematic therapy is medically indicated by the presence of at least one of the following:

A. >= 25 mucocutaneous (mouth or skin) lesions. B. Symptomatic visceral involvement. C. Symptomatic lymphedema (pain).

* Minimum of 5 clearly measurably cutaneous lesions by physical exam or measurable disease by X-ray, CT or MRI.
* Failed at least one systemic chemotherapy regimen.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Less than 2 weeks since major surgery.
* Serious uncontrolled infection. NOTE:
* Must be ruled out by thorough work-up in patients with unexplained fevers, night sweats, or involuntary weight loss of more than 10% normal weight.
* Leukopenia.
* Thrombocytopenia.

Patients with the following prior conditions are excluded:

* History of angina or myocardial infarction within the past 6 months.
* Second degree or third degree atrioventricular block without a pacemaker.
* Congestive heart failure (poorly controlled).
* History of prior malignancy except:

Completely excised in situ, carcinoma of the cervix or nonmelanomatous skin cancer.

Curatively treated other malignancy with no evidence of disease for at least 5 years.

Prior Medication:

Excluded:

Prior taxane therapy.

Required:

* At least one systemic chemotherapy regimen that failed to maintain significant benefit. NOTE:
* Intralesional chemotherapy regimens are not considered as prior chemotherapy.
* At least 2 weeks since last dose of prior systemic chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Gen Hosp / AIDS Oncology Research, Boston, Massachusetts, United States